CLINICAL TRIAL: NCT07100158
Title: The Diagnostic Value of Ultrasonographic Optic Nerve Sheath Diameter Measurement in Postdural Puncture Headache
Brief Title: Ultrasonographic Optic Nerve Sheath Diameter in Postdural Puncture Headache Diagnosis
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Other Study IDs: ONSD
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Anesthesia, Local; Headache
Keywords: Optic Nerve Sheath Diameter; Post-Dural Puncture Headache; Spinal Anesthesia
MeSH Terms: conditions — Headache; Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonographic Measurement of Optic Nerve Sheath Diameter (ONSD) — Non-invasive ultrasonographic measurement of optic nerve sheath diameter (ONSD) using a 7.5 MHz linear probe at predefined time points: preoperative and postoperative 6, 12, 24, 36, and 48 hours.

SUMMARY:
This study aims to investigate the hypothesis that ultrasonographic optic nerve sheath diameter (ONSD) measurement can help predict the development and severity of postdural puncture headache (PDPH) in patients undergoing spinal anesthesia for total knee arthroplasty. PDPH is defined as a headache that worsens in an upright position and improves while lying down.

DETAILED DESCRIPTION:
This prospective observational study aims to investigate the role of ultrasonographically measured optic nerve sheath diameter (ONSD) in predicting the development and severity of post-dural puncture headache (PDPH) in patients undergoing total knee arthroplasty (TKA) under spinal anesthesia.

The study will include patients aged 18 to 65 years, with American Society of Anesthesiologists (ASA) physical status I or II, who are scheduled to undergo total knee prosthesis (TKP) surgery under spinal anesthesia, with successful administration using a 27G Quincke spinal needle on the first attempt. Exclusion criteria will include a history of central nervous system disorders (e.g., cerebrovascular diseases, intracranial hemorrhage, brain tumors), ophthalmological disorders, hypertension, hepatic encephalopathy, renal failure, pregnancy, history of chronic headache or migraine, obesity (body mass index >35 kg/m²), alcohol or substance dependence, psychiatric disorders, local infection at the injection site, allergy to local anesthetics, bleeding diathesis, requirement for sedation during the procedure, conditions that may impair postoperative cooperation (e.g., mental retardation, language acquisition deficits), and inability to obtain reliable optic nerve sheath diameter (ONSD) measurements.

Ultrasonographic ONSD measurements will be performed using a 7.5 MHz linear ultrasound probe preoperatively (baseline) and at 6, 12, 24, 36, and 48 hours postoperatively. PDPH will be defined as a headache that worsens in the sitting or standing position and improves when lying down. Headache severity will be assessed using the Numerical Rating Scale (NRS), in which patients rate their pain from 0 (no pain) to 10 (the worst pain imaginable). Postoperative pain related to surgery will also be assessed using the NRS, and the need for rescue analgesics will be documented (NRS ≥ 4). Intraoperative vital parameters, including heart rate and arterial blood pressure, will also be monitored. In addition to the incidence and severity of PDPH, associated symptoms (nausea, vomiting, photophobia, diplopia, auditory symptoms, neck pain, and dizziness) will be recorded. Patients who develop PDPH will be assigned to Group H, while those who do not will be assigned to Group C.

The primary aim of this study is to determine the diagnostic and prognostic value of ONSD measurements in predicting PDPH following spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* ASA physical status I or II
* Scheduled for total knee arthroplasty under spinal anesthesia
* Successful spinal anesthesia with a single attempt using a 27G Quincke spinal needle
* Provided informed consent to participate in the study

Exclusion Criteria:

* History of neurological or central nervous system disorders (e.g., cerebrovascular disease, intracranial hemorrhage, brain tumor)
* Ophthalmological disorders
* Hypertension
* Hepatic encephalopathy
* Renal failure
* Pregnancy
* History of chronic headaches or migraine
* Obesity (BMI > 35 kg/m²)
* Alcohol or substance abuse
* Psychiatric disorders
* Local infection at the injection site
* Allergy to local anesthetics
* Bleeding diathesis
* Requirement for sedation during the procedure
* Inability to cooperate postoperatively (e.g., mental retardation, language deficits)
* Inability to obtain reliable ONSD measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years undergoing total knee arthroplasty under spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-Dural Puncture Headache (PDPH) | Within 48 hours postoperatively
  The proportion of patients who develop PDPH within the first 48 hours following spinal anesthesia. PDPH will be defined as a headache that worsens in the sitting or standing position and improves when lying down.

SECONDARY OUTCOMES:
Optic Nerve Sheath Diameter (ONSD) Measurement | At baseline (preoperative), and at 6, 12, 24, 36, and 48 hours postoperatively
  ONSD will be measured via ultrasonography using a 7.5 MHz linear probe placed over the closed upper eyelid with a thin layer of gel. Two measurements will be obtained in transverse and sagittal planes for each eye, and the average of four measurements will be recorded as the final ONSD value.
Severity of Post-Dural Puncture Headache (PDPH) | Within 48 hours postoperatively
  Headache severity will be assessed using the 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst possible pain. Assessments will be conducted in patients who develop PDPH.
Symptoms Associated with PDPH | Within 48 hours postoperatively
  Presence of associated symptoms such as nausea, vomiting, photophobia, diplopia, hearing disturbances, neck pain, and dizziness will be recorded in patients diagnosed with PDPH. Symptoms will be defined based on patient reports and clinical assessment
Postoperative Pain | Within 48 hours postoperatively
  Pain at the surgical site will be assessed using the 11-point Numerical Rating Scale (NRS), where 0 indicates "no pain" and 10 indicates "the worst pain imaginable." Pain scores will be recorded regardless of the presence of PDPH.
Rescue Analgesic Requirement | Within 48 hours postoperatively
  Patients with postoperative pain scored 4 or higher on the 0-10 Numerical Rating Scale (NRS) will receive 100 mg of intravenous tramadol as rescue analgesia. The total number of administered rescue analgesic doses will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No